CLINICAL TRIAL: NCT03268733
Title: The Clinical and Biochemical Effects of Folic Acid on Sudanese Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: The Effects of Folic Acid on Sudanese Women With Polycystic Ovary Syndrome
Acronym: FolicacidPCOS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Khartoum (Other)
Collaborators: Awad, Mohamed Ibrahim, M.D. (Individual); Duria abdulwahab Elrrayes (Unknown)
Responsible Party: Principal Investigator, Mohammed Hassan Alnazeer, Clinical Pharmacist, University of Khartoum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Folic acid in PCOS
Record Dates: First submitted 2017-08-24; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Folic acid; PCOS; Insulin resistance; Infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Infertility | interventions — Folic Acid

STUDY DESIGN:
Intervention Model Description: Open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): 45 PCOS patients will receive 5 mg folic acid
  Interventions: Drug: Folic Acid
- control group (No Intervention): 45 PCOS patients will receive no folic acid

INTERVENTIONS:
Drug: Folic Acid — Tablet 5 mg
  Arms: Treatment group

SUMMARY:
An open clinical trial

DETAILED DESCRIPTION:
The patients with PCOS will be recruited to receive folic acid (45 patients) and equal number will receive no folic acid

ELIGIBILITY:
Inclusion Criteria:

* Patients who will visit this centre suffering from PCOS-related subfertility will be invited to be enrolled to this study if met the Rotterdam criteria for the diagnosis of PCOS

Exclusion Criteria:

* The patients whom will be excluded from the study are those comorbid with hyperprolactinemia, congenital adrenal hyperplasia, diabetes mellitus, significant cardiovascular problems, thyroid dysfunctions, unresolved medical conditions, or using medications suspected to affect reproductive or metabolic functions within two months of the study entry.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female patients suffering from PCOS-related subfertility
Enrollment: 90 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
pregnancy rates | 3 months
  Pregnancy rates will be compared in the treatment group and control group
Ovulatory pattern improvements | 3 months
  Ovulatory pattern will be assessed based on the history of the PCOS patients, the patients whom were having baseline oligomenorrhea or amenorrhea will be re-assessed for resuming regular cycles defined as periods lasting 22 - 35 days. this pattern improvement will be compared in the treatment group and control group using questionnaire
Clinical signs of hyperandrogenemia | 3 months
  Hirsutism will be used as a sign of hyperandrogenemia, Patients will be provided with modified Ferriman -Gallwey (mFG) images to self-rate hair growth in each of the 9 body areas (upper lip, chin, chest, upper and lower back, upper and lower abdomen, thighs, and upper arms). For each site, a score on a scale of 0 to 4 was recorded. A total score of 8 or greater is defined as clinical evidence of hirsutism; scores from 8 to 15 are considered mild hirsutism; scores from16 to 25 are considered moderate; and scores from 26 to 36 are considered severe hirsutism. The baseline and after 3 months hirsutism compared in the treatment group and control group

SECONDARY OUTCOMES:
Plasma level of testosterone | 3 months
  Plasma level of testosterone will be compared in the treatment group and control group
Plasma level of insulin | 3 months
  Plasma level of insulin will be compared in the treatment group and control group
Plasma level of follicle-stimulating hormone (FSH) | 3 months
  Plasma level of follicle-stimulating hormone will be compared in the treatment group and control group
Plasma level of luteinizing hormone (LH) | 3 months
  Plasma level of luteinizing hormone will be compared in the treatment group and control group

OTHER OUTCOMES:
Lipid profile | 3 months
  Lipid profile will be compared in the treatment group and control group
Plasma level of random glucose | 3 months
  Plasma level of random glucose will be compared in the treatment group and control group
Plasma level of folate | 3 months
  Plasma level of folate will be compared in the treatment group and control group
Plasma level of homocysteine (Hcy) | 3 months
  Plasma level of homocysteine (Hcy) will be compared in the treatment group and control group
Plasma level of hemoglobin (Hb) | 3 months
  Plasma level of hemoglobin (Hb) will be compared in the treatment group and control group
Plasma level of C-reactive protein (CRP) | 3 months
  Plasma level of C-reactive protein (CRP) will be compared in the treatment group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Hassan Alnazeer, Study Chair — University of Khartoum
Locations (1):
- Saad Abul ella fertility Centre, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Undecided
still undecided